CLINICAL TRIAL: NCT07298044
Title: A Prospective, Single-arm, Phase 4 Study to Evaluate the Course of Serum Transthyretin (TTR) Level With Acoramidis in Adult Patients With Variant or Wild-type Transthyretin Amyloidosis With Cardiomyopathy (ATTR-CM) Previously Treated With Tafamidis
Brief Title: A Study to Learn More About the Change in the Blood Levels of Transthyretin When Participants With Transthyretin Amyloidosis With Cardiomyopathy Switch From Tafamidis to Acoramidis
Acronym: ACO-SWITCH
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23026
Record Dates: First submitted 2025-12-11; First posted 2025-12-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Transthyretin Amyloid Cardiomyopathy
Keywords: ATTR-CM
MeSH Terms: interventions — attruby

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acoramidis (Experimental): Participants will receive acoramidis 712 mg orally BID
  Interventions: Drug: Acoramidis

INTERVENTIONS:
Drug: Acoramidis — 356 mg film-coated tablets.
  The recommended dose of acoramidis is 712 mg (two tablets, 356 mg) orally, twice daily, corresponding to a total daily dose of 1424 mg.
  Other Names: BAY3684938, BEYONTTRA

SUMMARY:
Transthyretin (TTR) is a protein made by the liver that helps transport thyroid hormone and vitamin A in the blood. In some people, this protein breaks down and forms harmful clumps called amyloid. TTR amyloid gets deposited in the heart wall and stops it from pumping blood properly, which may lead to heart failure. The breakage in TTR protein can be age-related (wild-type ATTR-CM), or genetic (variant ATTR-CM).

The study drug, acoramidis, works by attaching itself to the TTR protein, making TTR more stable and less likely to break down and form amyloid (clumps). This helps to slow down the progression of the disease, improve heart function, and increase the TTR levels in the blood. Acoramidis is an approved treatment for wild-type or variant ATTR-CM in Europe and the United States.

Tafamidis is another drug that stabilizes TTR and prevents it from breaking down.

In this study, acoramidis will be studied in participants with ATTR--CM who were previously treated with tafamidis. The main purpose of this study is to assess the change in blood TTR levels after participants are switched from tafamidis to acoramidis. This will be studied to understand if acoramidis causes an increase in blood TTR levels beyond the levels achieved with tafamidis.

For this, the researchers will measure the change in the levels of TTR protein in participants' blood after 6 months of the treatment with acoramidis, or earlier if a participant stops the treatment before reaching that six-month mark.

All participants will continue taking tafamidis during the screening period. In the treatment period of the study, participants will take acoramidis as two tablets twice daily by mouth, for up to 6 months.

At the start of this study, the study doctors will review each participant's medical history and check their overall health. The study doctors will perform electrocardiograms (ECG), and measure blood pressure and heart rate. Researchers will also take blood and urine samples from the participants to measure levels of TTr, NT-proBNP, hs-TnT, hs-CRP, RBP4, eGFR, creatinine, cystatin-C, UACR, and TSH at the start of the study, and at various time points thereafter (during the study) to assess heart, kidney and thyroid function.

There will be a total of 9 study check-ins. Participants will visit the study site twice: at screening and at the end of treatment period. A study nurse will visit the participant's home 6 times, at the start of treatment, Weeks 1, 2, 3 and 4, then again at 3 months. The final check-in will be done by phone.

The study doctors will monitor the health of the participants regularly for any medical problems during follow-up visits. Participants will know the treatment they will receive during the study. Each participant could be in the study for about 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 to 90 years of age inclusive, at the time of signing the informed consent.
* Diagnosis of ATTR-CM; disease defining examination, i.e., Single Photon Emission Computed Tomography (SPECT) or SPECT/Computed Tomography (CT) or biopsy, within 24 months prior to Visit 1 (V1).
* Participants must currently be treated with tafamidis and have used tafamidis for at least the previous 3 months prior to V1 and have adhered to tafamidis therapy.
* New York Heart Association (NYHA) class ≤ II at V1.
* Estimate glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73m^2 at V1.
* N-terminal pro-B-type Natriuretic Peptide (NT-proBNP) > 300 and ≤ 7000 pg/mL at V1.

Exclusion Criteria:

* Prior liver or heart transplantation or planned within the next 12 months.
* Current or planned use of ventricular assist device.
* Active cancer or other disease that decreases the life expectancy to less than one year.
* Heart failure due to ischemic heart disease.
* Myocardial infarction, cardiovascular (CV) surgery, or unstable angina within the last 90 days prior to V1.
* Confirmed diagnosis of light-chain amyloidosis.
* Dialysis or severe renal impairment as reflected by Urinary Albumin Creatinine Ratio (UACR) > 300 mg/g at V1.
* Major surgery 90 days prior to V1.
* Recent initiation of Sodium-Glucose-Cotransporter-2 inhibitors (SGLT2i) within 3 months before V1.
* Initiation of treatment with a diuretic or increase in diuretic dose within 3 months before V1.
* Treatment with calcium channel blockers (e.g., verapamil, diltiazem) or digitalis.
* Recent CV hospitalization within 3 months before V1.
* Known hypersensitivity to acoramidis or to any of the excipients.
* A condition that, as judged by the investigator, would preclude compliance with the study protocol, such as a history of substance abuse, alcoholism, or a psychiatric condition.
* Known or suspected liver disorder and bile secretion/flow (cholestasis, also history of it).
* Abnormal liver function tests at V1, defined as ALT (GPT) or AST (GOT) ≥ 3 x ULN or total bilirubin ≥ 3 x ULN at V1.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-13 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in serum TTR level from baseline to month 6 or premature discontinuation of treatment | From baseline to month 6 or premature discontinuation of treatment
  TTR = Transthyretin

SECONDARY OUTCOMES:
Serum TTR level at baseline, week 1, 2, 3, 4 and at month 3. | At baseline, week 1, 2, 3, 4 and at month 3
  TTR = Transthyretin
Number of participants with TEAEs and serious TEAEs | From the first administration of study drug until 30 days after the last dose of study drug or end of study, whatever occurs first
Change from baseline to month 6 of NT-proBNP | From baseline to month 6
  NT-proBNP = N-terminal pro-B-type Natriuretic Peptide
Change from baseline to month 6 of hs-TnT | From baseline to month 6
  hs-TNT = high-sensitivity Troponin T
Change from baseline to month 6 of hs-CRP | From baseline to month 6
  hs-CRP = high-sensitivity C-reactive protein
Change from baseline to month 6 of RBP4 | From baseline to month 6
  RBP4 = Retinol Binding Protein 4
Signs of cardiac remodeling from baseline to month 6 | From baseline to month 6
  These signs will be measured by echocardiogram
Change from baseline to month 6 in 6MWD | From baseline to month 6
  The 6-Minute Walk distance (6MWD) measures the total distance that a participant could walk in 6 minutes.
Change from baseline to month 6 in the eGFR | From baseline to month 6
  eGFR = estimated glomerular filtration rate
Change from baseline to month 6 in Creatinine | From baseline to month 6
Change from baseline to month 6 in Cystatin C | From baseline to month 6
Change from baseline to month 6 in UACR | From baseline to month 6
  UACR = Urinary Albumin Creatinine Ratio
Change from baseline to month 6 in TSH | From baseline to month 6
  TSH = Thyroid Stimulating Hormone
Change from baseline to month 6 in KCCQ-OS score | From baseline to month 6
  The Kansas City Cardiomyopathy Questionnaire-Overall Summary (KCCQ-OS) is 23-item questionnaire developed to measure health status and health-related quality of life (QoL) in individuals with heart failure. Items include heart failure symptoms, impact on physical and social functions, and how heart failure impacts QoL.
Change from baseline to month 6 of EQ-5D-5L index score | From baseline to month 6
  The EuroQol-5-Dimension-5-Level (EQ-5D-5L) includes two parts. In the first part, participants are asked to rate their current health state on 5 dimensions (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with each dimension having five levels of function (1-no problem, 2-slight problem, 3-moderate problem, 4-severe problem, and 5-extreme problem). The second part is a self-rating of current health status on a Visual Analogue Scale (EQ VAS) with endpoints labeled "best imaginable health state" (score of 100) and "worst imaginable health state" (score of 0). The scores from the 5 dimensions are used to calculate the index score.

CONTACTS AND LOCATIONS:
Locations (5):
- Austria (5):
  - Universitätsklinikum St. Pölten - Lilienfeld - Klinische Abteilung für Innere Medizin 3, Sankt Pölten, Lower Austria
  - Medizinische Universität Graz- Klinische Abteilung für Kardiologie, Vienna, Styria
  - Medizinische Universität Wien- Universitätsklinik für Innere Medizin II, Klinische Abteilung für Kardiologie, Vienna, Vienna
  - Klinik Favoriten - 5.Medizinische Abteilung-Kardiologie, Vienna, Vienna
  - Klinik Ottakring - 3. Medizinische Abteilung mit Kardiologie, internistischer Intensivmedizin und Ambulanz, Vienna, Vienna

IPD SHARING:
Plan to Share IPD: No
Currently, there is no established plan for the sharing of Individual Patient Data (IPD) from this study. The availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA 'Principles for responsible clinical trial data sharing.' This pertains to the scope, timepoint, and process of data access.
  As such, Bayer commits to considering requests from qualified researchers for patient- / study-level clinical trial data, and documents from clinical trials involving medicines and indications approved in the US and EU. However, this commitment does not reflect an active IPD sharing plan. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Researchers can use www.vivli.org to request access to IPD and documents from clinical studies to conduct research. Information on Bayer's criteria for listing studies is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/23026